CLINICAL TRIAL: NCT03910140
Title: A Prospective Non-controlled Single-arm Study of TILA-TACE in Treatment of Hepatocellular Carcinoma
Brief Title: TILA-TACE in Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZUSAHZUCI201701
Record Dates: First submitted 2019-02-18; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Tumor Response Rate; Overall Survival
MeSH Terms: interventions — Radiotherapy, Conformal; Sirtuins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TILA-TACE group (Experimental)
  Interventions: Procedure: TILA-TACE treatment

INTERVENTIONS:
Procedure: TILA-TACE treatment — TACE was performed through the transfemoral route using a 5-Fr catheter (Shepherd-hook modified Angiographic Catheter, HANACO Medical, Tian Jin, China ) that was advanced from celiac artery to common hepatic artery, proper hepatic artery, hepatic artery and ultimately to tumor feeding arteries which are defined by angiography. Then, a coaxial microcatheter (2.8 Fr Marguerite II, ASAHI INTECC GMA CO., LTD, Nagoya, Japan) was selectively inserted through a 5-Fr catheter into the tumor feeding artery, into which, 5% sodium bicarbonate was infused alternatively with doxorubicin-lipiodol emulsion. Finally, the artery was embolized with PVA (Embosphere®, BioSphere Medical, Paris, France) and microcoil ( Tornado ®, COOK Medical, USA).
  Other Names: 3D-CRT; SBRT; SIRT

SUMMARY:
To validate the tumor response rate: in the previous study, the investigators showed that TILA-TACE achieved 100% tumor response rate. However, as the study sample size was 40, the investigators need to validate the tumor response rate using a larger sample size; To validate the overall survival: in the previous study, the investigators showed that TILA-TACE significantly prolonged the overall survival of the patients with large and massive tumor. Again, the sample size was small, the investigators need to validate the data using a large sample size.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma is confirmed by tissue pathology or in accordance with clinical diagnosis standard;
* ECOG score 0-1;
* HCC BCLC grading 0, A, B, C;
* Child-Pugh score prior to therapy A and B;
* As judged by investigators, the patient can comply with the study protocol;
* Patient voluntarily participates in this study, understands the process of the study, and is willing to sign the written consent form.

Exclusion Criteria:

* HCC BCLC grading D;
* Child-Pugh score prior to therapy C.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The response to treatment | 1 month after therapy
  Viable tumors were assessed by MRI according to EASL criteria. The enhanced and non-enhanced areas represent viable and necrotic tumors. At least 2 radiologists evaluate the approximate viable tumor residues (%) of total tumor volume (Total tumor volume was the sum of viable and necrotic volume).
  The response to treatment is defined by the Viable Tumor Residues (%) as below: complete response (CR), no obvious viable residuals; near complete response (NCR), viable residuals <10%; partial response (PR), viable residuals >10% but < 50%; stable disease (SD), viable tumor residuals between >50% but ≤100%; and progressive disease (PD), viable tumors > 100%.

SECONDARY OUTCOMES:
Lifetime (months) | 6 months once after therapy
  Record the survival time of patients by follow up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
share data for several times in experiment; Research Manager: http://www.medresman.org/login.aspx